CLINICAL TRIAL: NCT07011459
Title: Community Teaching Kitchen-based Culinary Education as a 'Food is Medicine' Solution for Improving Health Equity Among Racially/Ethnically Diverse Seniors
Brief Title: The Cooking for Health Optimization and Disease Prevention (CHOP) Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: Humana Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-1940
Record Dates: First submitted 2025-05-16; First posted 2025-06-08 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular Diseases
Keywords: Culinary; Cardiometabolic health; Mental health; Mediterranean Diet; Nutrition
MeSH Terms: conditions — Cardiovascular Diseases; Psychological Well-Being | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culinary intervention group (Active Comparator): The interventions include the teaching-kitchen based structured, hands-on culinary education classes.
  Interventions: Behavioral: Cooking class
- Usual diet control group (Placebo Comparator): Participants randomized to the usual diet group will not receive culinary education classes, while they will continue to receive clinical care recommendations from their physician(s).
  Interventions: Other: Standard of care

INTERVENTIONS:
Behavioral: Cooking class — 3-month community teaching kitchen-based culinary education of MedDiet
  Arms: Culinary intervention group
Other: Standard of care — Participants will continue to receive clinical care recommendations from their physicians
  Arms: Usual diet control group

SUMMARY:
Poor nutrition-related diseases disproportionately impact seniors and racial/ethnic minorities who are more likely to experience disparities in proper nutrition. Culinary medicine is a new evidence-based educational approach that blends the art of food and cooking with the science of medicine. Recently, culinary medicine is proposed by the 2020-2030 Strategic Plan for NIH Nutrition Research and national 'Food is Medicine (FIM)' Movement as potential solutions for improving healthy eating, creating social and emotional connections, and nutrition-related health equity. Built upon the well-established community teaching kitchen at The Goldring Center for Culinary Medicine (GCCM) at Tulane University and nearly 10 years of experience in delivering culinary education of Mediterranean diet (MedDiet), the investigators will conduct a randomized controlled trial (RCT) to test the feasibility and effectiveness of 3-month community teaching kitchen-based culinary education of MedDiet on improving cardiometabolic and mental health among racially and ethnically diverse seniors.

DETAILED DESCRIPTION:
The study is designed as a two-arm parallel-group randomized controlled trial (RCT). The interventions in the two groups are described as below:

i) Culinary intervention group (n=48): The interventions include the teaching-kitchen based structured, hands-on culinary education classes.

ii) Usual diet control group (n=48): Participants randomized to the usual diet group will not receive culinary education classes, while they will continue to receive clinical care recommendations from their physician(s).

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years or older
* English speaking
* Ability to provide informed consent.

Exclusion Criteria:

* Medical history of cardiovascular disease (CVD) or cancer.
* Food allergies including, but not limited to, milk, eggs, shellfish, nuts, wheat or gluten, and soy.
* Special diets including, but not limited to, Mediterranean, veganism, vegetarianism, gluten-free, and the ketogenic diet.
* Current use of medications that could affect blood glucose and lipids levels including, but not limited to, insulins (Humalog, Novolog, insulin detemir, etc.), anti-diabetic medications (metformin, sulfonylureas, meglitinides, etc.), Ozempic. HAART, and beta blockers.
* No children are involved.
* No other vulnerable subjects will be involved.

Ages: 55 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in blood pressure measurements | Baseline, 3 months
  The investigators will measure the change in blood pressure from baseline visit 1 to visit 3. The average of 3 blood pressure readings will be taken. They will be measured at baseline visit and at 3 months visit.
Change in blood glucose measurements | Baseline, 3 months
  The investigators will measure the change in blood glucose. The fasting blood glucose will be measured at baseline and at 3 months visit. A continuous glucose monitoring (CGM) device will be used as well to measure the change in blood glucose.
Change in blood lipid profile measurements | Baseline, 3 months
  The investigators will measure the change in blood lipid profile. The blood lipid profile will be measured at baseline and at 3 months visit.

SECONDARY OUTCOMES:
Change in cognitive function measured using the Montreal Cognitive Assessment (MoCA) | Baseline, 3 months
  The investigators will measure the change in cognitive function using the Montreal Cognitive Assessment. It is a screening tool used to assess cognitive function. A higher score indicates less severe cognitive impairment. The grading scale for the MoCA is as follows:
  0-9: Severe cognitive impairment 10-17: Moderate cognitive impairment 18-25: Mild cognitive impairment 26-30: Normal cognitive function
  This will be measured at baseline visit and at 3 months visit.
Depression severity assessment using the PHQ-9 (Patient Health Questionnaire) | Baseline, 3 months
  The investigators will assess the depression severity using the PHQ-9 (Patient Health Questionnaire) It is a self-reporting scoring system which assigns points to each question based on the frequency of reported symptoms, with a total score ranging from 0 to 27. The total score can then be used to determine the possible level of depression severity. The higher the score, the more severe depression level will be.
  0-4 points: None to minimal depression. 5-9 points: Mild depression. 10-14 points: Moderate depression. 15-19 points: Moderately severe depression. 20-27 points: Severe depression.
  This will be measured at baseline visit and at 3 months visit.
Loneliness severity assessment using the UCLA Loneliness Scale Version 3 (UCLA-LS) | Baseline, 3 months
  The investigators will assess the loneliness severity using the UCLA Loneliness Scale Version 3 (UCLA-LS). It is a self-reporting questionnaire used to measure an individual's feelings of loneliness. It's scored by combining the total of responses to 20 questions, where higher scores generally indicate greater feelings of loneliness. The interpretation of scores often uses a categorization based on the total score, with scores above 43 generally indicating a high degree of loneliness.
  Low Loneliness: Total score < 28. Moderate Loneliness: Total score 28-43. High Loneliness: Total score > 43.
  This will be measured at baseline visit and at 3 months visit.
Social Anxiety Disorder assessment using the Severity Measure for Social Anxiety Disorder (Social Phobia Scale for Adults) questionnaire | Baseline, 3 months
  The investigators will assess Social Anxiety Disorder using the Severity Measure for Social Anxiety Disorder (Social Phobia Scale for Adults). It is a 10-item questionnaire, used to assess social anxiety (social phobia) in adults.
  Total Score Range: 0-40. Interpretation: Higher scores correlate with more severe social phobia symptoms.
  Cut-off Score: 24 or above may indicate a presence of non-generalized social phobia.
  This will be measured at baseline visit and at 3 months visit.
Mediterranean eating pattern assessment using the Mediterranean Diet Adherence Screener (MEDAS) questionnaire | Baseline, 3 months
  The investigators will assess the Mediterranean eating pattern using the Mediterranean Diet Adherence Screener (MEDAS) questionnaire. It is used to assess how someone's diet aligns with a traditional Mediterranean eating pattern. A higher score means better adherence.
  0-4 points: Generally considered low adherence. 5-9 points: Considered moderate to fair adherence. 10-14 points: Indicates good or very good adherence.
  This will be measured at baseline visit and at 3 months visit.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Qi, PhD, MD, Principal Investigator — Tulane University
Locations (2):
- United States (2):
  - The Goldring Center for Culinary Medicine, New Orleans, Louisiana
  - Tulane Weatherhead School of Public Health and Tropical Medicine, New Orleans, Louisiana